CLINICAL TRIAL: NCT03967106
Title: Role of Remote Ischaemic Preconditioning on Activity, Fatigue and Gait in People With Multiple Sclerosis.
Brief Title: RIPC on Activity, Fatigue and Gait in MS
Acronym: MSIPC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: JP Moulton Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STH20727
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: remote ischaemic preconditioning; gait analysis; activity; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue | interventions — Ischemic Preconditioning; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either the treatment or sham condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischaemic preconditioning (Experimental): Remote IPC (RIPC) intervention daily for six weeks.
  Interventions: Other: Ischaemic Preconditioning
- Sham (Sham Comparator): Remote sham intervention daily for six weeks.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Ischaemic Preconditioning — IPC to the upper arm using a manual blood pressure machine with cuff. Three cycles of 5 minute cuff inflation to 30mmHg above the systolic blood pressure (BP) followed by 5 minute cuff deflation.
  Arms: Remote Ischaemic preconditioning
Other: Sham — Sham intervention to the upper arm using a manual blood pressure machine with cuff. Three cycles of 5 minute cuff inflation to 30mmHg below the diastolic blood pressure (BP) followed by 5 minute cuff deflation.
  Arms: Sham

SUMMARY:
This study evaluates whether Remote Ischaemic Preconditioning (RIPC) can improve activity, gait and fatigue in people with Multiple Sclerosis. Half the participants will receive RIPC, the other half will receive a sham treatment.

DETAILED DESCRIPTION:
Regular physical activity has been shown to improve physical fitness, fatigue, quality of life, and reduce the progression of disability in people with multiple sclerosis (MS). However, people with MS are less physically active than others. This is partly due to poor exercise tolerance and fatigue.

Remote Ischemic preconditioning (RIPC) is the exposure of a limb to brief periods of circulatory occlusion and reperfusion by inflating pressure cuffs around arms or legs to above systolic pressures (mmHg), to protect organs against ischaemic injury. RIPC has been shown to improve exercise performance and delay fatigue in athletes. However, there is little to no research examining the effect of RIPC on walking or exercise performance in MS patients. The aim of this trial is to assess whether RIPC can improve activity, gait and reduce fatigue in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as per the McDonald's criteria
* Sufficient cognitive ability and understanding of the English language to give informed consent and complete study questionnaires
* Ability to walk for 6 minutes without rest
* Resting Systolic BP of more than 100mmHg
* Resting Systolic BP of less than 170mmHg

Exclusion Criteria:

* Cognitive difficulties or insufficient English to allow understanding of consent and study questionnaires
* Inability to walk
* Other systemic illness affecting exercise tolerance
* Resting Systolic BP of less than 100mmHg
* Resting systolic BP of 170mmHg or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in speed of walking over a one week period | 7 weeks
  Change in activity levels will be assessed by measuring the average speed of participants walking during the waking hours over a one week period, using a wearable activity monitor for one week before the intervention and during the final week of the 6 week intervention period.
Change from baseline in number of steps taken over a one week period | 7 weeks
  Change in activity levels will be assessed by measuring the average number of steps taken during the waking hours over a one week period, using a wearable activity monitor for one week before the intervention and during the final week of the 6 week intervention period.
Change from baseline in length of stride over a one week period | 7 weeks
  Change in activity levels will be assessed by measuring the average length of stride during the waking hours over a one week period, using a wearable activity monitor for one week before the intervention and during the final week of the 6 week intervention period.
Change from baseline in speed of walking during the 6 minute walk test | 6 weeks
  Speed of walking during the 6 minute walk test will be assessed using wearable sensors at baseline and after the 6 week intervention period. The 6 minute walk test assesses exercise tolerance by assessing walking over the span of six minute.
Change from baseline in Modified Fatigue Impact Scale (MFIS) Score | 6 weeks
  A 21 item self reported fatigue scale which assess the effects of fatigue across three domains, cognitive, physical and psycho-social. Each item is scored from 0-4 (0=no effect of fatigue, 4=large effect of fatigue) yielding a total between 0 - 84.
Change from baseline in Multiple Sclerosis Walking Scale 12 (MSWS-12) score | 6 weeks
  A 12 item self reported scale which assesses the impact of MS on a patient's walking ability. Each item is scored from 1-5 (1=no impact, 5=high impact), yielding a total between 1-60 which is transformed to a percentage out of 100.
Change from baseline in Borgs rating of perceived exertion scale score | 6 weeks
  Exertion after the 6 minute walk test will be measured at baseline and following the 6 week intervention period using the Borgs rating of perceived exertion scale, a self report measure of perceived exertion ranging from 6-20 (6=no exertion, 20=exhaustion).

CONTACTS AND LOCATIONS:
Overall Officials: Siva Nair, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided